CLINICAL TRIAL: NCT07017790
Title: Amino Acid PET Imaging to Assess the Efficacy of IDH Inhibitor Treatments for Patients With Refractory IDH Mutated Gliomas
Brief Title: Amino Acid PET to Assess the Efficacy of IDH Inhibitor Treatments for IDH Mutated Gliomas
Acronym: TEP-IDH
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, Principal investigator, Central Hospital, Nancy, France
Other Study IDs: 2025PI093
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Amino-acid PET — Patients received 18-fluoroDopa then a PET exam

SUMMARY:
Amino acid PET imaging could represent a biomarker for the evaluation of IDH inhibitor treatments for patients with refractory IDH-mutated gliomas

DETAILED DESCRIPTION:
Amino acid PET imaging could represent a biomarker for the evaluation of IDH inhibitor treatments for patients with refractory IDH-mutated gliomas In fact, this study will allow us to assess, using Rano 1.0 criteria for PET and Rano 2.0 criteria for MRI, which of the two examinations is most effective in assessing the efficacy of anti-IDH treatment patients with refractory IDH-mutated gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent amino acid PET for early assessment of therapeutic response of IDH-mutated gliomas under anti-IDH treatment between February 2022 and November 2024

Exclusion Criteria:

* Individuals who have objected to the use of their data

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent amino acid PET for early assessment of therapeutic response of IDH-mutated gliomas under anti-IDH treatment between February 2022 and November 2024
Sampling Method: Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Compare the performance between amino acid PET and brain MRI to assess a treatment efficacy | one day
  Comparison between early therapeutic response according to RANO 1.0 and RANO 2.0 PET criteria and tumor progression at 6 months

SECONDARY OUTCOMES:
Compare the performance between amino acid PET and brain MRI to assess a treatment efficacy for the identification of lesions | one day
  Determination of the number of lesions assessable by amino acid PET according to RANO 1.0 PET criteria and by MRI according to RANO 2.0 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU of NANCY, Vandœuvre-lès-Nancy, France